CLINICAL TRIAL: NCT01971658
Title: A PHASE III STUDY OF VELCADE (BORTEZOMIB) THALIDOMIDE DEXAMETHASONE (VTD) VERSUS VELCADE (BORTEZOMIB) CYCLOPHOSPHAMIDE DEXAMETHASONE (VCD) AS AN INDUCTION TREATMENT PRIOR TO AUTOLOGOUS STEM CELL TRANSPLANTATION IN PATIENTS WITH NEWLY DIAGNOSED MULTIPLE MYELOMA."
Brief Title: Efficacy Study Comparing Velcade Dexamethasone Thalidomide Versus Velcade Cyclophosphamide Dexamethasone as Induction Treatment in the Initial Management of Multiple Myeloma (IFM2013-04)
Acronym: IFM2013-04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC13_0284; 2013-003174-27 (EudraCT Number)
Record Dates: First submitted 2013-09-30; First posted 2013-10-29 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Newly Diagnosed
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Cyclophosphamide; Bortezomib; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VELCADE (BORTEZOMIB) THALIDOMIDE DEXAMETHASONE (VTD) (Active Comparator): Arm A:
  1. Induction therapy 4 cycles of VTD (21 days) Thalidomide® 100 mg/day Per Os Day1 to Day21 Velcade® 1.3 mg/m²/day Subcutaneous Day1, 4, 8 and 11 Dexamethasone 40 mg/day Per Os Day 1 to 4 and Day 9 to 12
  2. Systematic stem cell harvest after cycle 3 Mobilization: Cyclophosphamide and one week after the last dose of Thalidomide, stem cells have to be harvested
  Interventions: Drug: Thalidomide®; Drug: Velcade®; Drug: Dexaméthasone
- VELCADE (BORTEZOMIB) CYCLOPHOSPHAMIDE DEXAMETHASONE (VCD) (Active Comparator): For arm B:
  1. Induction therapy : 4 cycles of VCD (21 days)
     * Cyclophosphamide 500 mg/m²/day, Per Os Day 1, 8, 15
     * Velcade® and Dexamethasone identical treatment to Arm A
  2. Systematic stem cell harvest after cycle 3 Mobilization: Cyclophosphamide and two weeks after the last dose of Cyclophosphamide, stem cells have to be harvested
  Interventions: Drug: Cyclophosphamide; Drug: Velcade®; Drug: Dexaméthasone

INTERVENTIONS:
Drug: Thalidomide®
  Arms: VELCADE (BORTEZOMIB) THALIDOMIDE DEXAMETHASONE (VTD)
Drug: Cyclophosphamide
  Arms: VELCADE (BORTEZOMIB) CYCLOPHOSPHAMIDE DEXAMETHASONE (VCD)
Drug: Velcade®
Drug: Dexaméthasone

SUMMARY:
This is a phase III, multicenter, prospective with a clinical benefit, open-label and randomized study to compare two different treatments : Velcade (Bortezomib) Thalidomide Dexamethasone (VTD) versus Velcade (Bortezomib) Cyclophosphamide Dexamethasone (VCD) as an Induction Treatment prior to Autologous Stem Cell Transplantation in patients with Newly Diagnosed Multiple Myeloma.

Eligible patients will be randomized into 2 treatment arms. Each patient will receive 4 consecutive 21 day cycles of an induction treatment with either VTD or VCD.

DETAILED DESCRIPTION:
The patient population will consist of adult men and women who have a confirmed diagnosis of Multiple Myeloma and who meet eligibility criteria. They will be recruited from among the patients consulting in an investigating centre's haematology service for newly diagnosed, symptomatic, untreated multiple myeloma.

in each treatment arm there will be :

1. Induction therapy : 4 cycles of VTD (21 days)or VCD
2. Systematic stem cell harvest after cycle 3

ELIGIBILITY:
Inclusion Criteria:

Patients newly diagnosed with symptomatic Multiple Myeloma (MM) patient

1. - 18 ≤ age < 66 years
2. - Eastern Cooperative Oncology Group Performance Status of 0, 1 or 2
3. - Patients must be eligible for Autologous Stem Cell Transplantation
4. - Patients must have measurable disease by serum M-protein ≥ 10 g/L and/or urine M-protein ≥200mg/day
5. - Female patients of child-bearing potential (FCBP):

   * Must agree to have medically supervised pregnancy tests prior to starting study and every 21 days, including 4 weeks after the end of study treatment. This applies even if the patient practices complete and continued sexual abstinence.
   * Must agree to use and be able to comply with effective contraception without interruption, 28 days prior to starting study drug, during the study therapy (including during periods of dose interruptions), and for 28 days after discontinuation of study therapy.
6. - Male Patients:

   * Must agree to use a condom during sexual contact with a FCBP, throughout study drug therapy, during any dose interruption and for one week after discontinuation of study therapy
   * Must agree to not donate semen during study drug therapy and for one week after discontinuation of study therapy
7. - All patients must:

   * Agree to abstain from donating blood while taking study drug therapy and for one week after discontinuation of study drug therapy
   * Agree not to share study medication with another person.
8. - Patients must be capable of giving informed consent
9. - Patients must be affiliated with French social security system

Exclusion Criteria:

1. - Asymptomatic Multiple myeloma
2. - Non-secretory Multiple myeloma
3. - Proven AL-amyloidosis
4. - Age ≥ 66 years old
5. - Prior or current systemic therapy for Multiple myeloma, including steroids (except for emergency use of a 4-day block of dexamethasone before randomization, maximum total dose allowed 160 mg)
6. - Radiation therapy in the 2 weeks preceding randomization
7. - National Cancer Institute grade ≥ 2 peripheral neuropathy
8. - Haemoglobin < 8g/dL
9. - Absolute neutrophil count < 1,000 cells / µL, platelet count < 50,000 cells / µL
10. - Creatinine level > 170 µmol/L or requiring dialysis.
11. - Bilirubin, transaminases or GamaGT > 3 UNL (upper normal limit)
12. - Positive HIV serology, evidence of active Hepatitis B and C infection
13. - Severe active infection
14. - Inability to comply with an anti-thrombotic treatment regimen
15. - A personal medical history of severe psychiatric disease
16. - Uncontrolled diabetes contraindicating the use of high-dose dexamethasone
17. - Non-controlled or severe cardiovascular disease (including a myocardial infarction in the 6 months prior to recruitment)
18. - A personal medical history of cancer unless the patient has been without relapse after treatment discontinuation > or = 5 years (except for basocellular skin cancer or in situ cervical cancer)
19. - Use of any investigational drug in the 30 days preceding randomization

22 - Pregnant or lactating women. 23 - Adults under juridical protection 24 - Known or suspected hypersensitivity to any of the study therapies or excipients 25 - Necessity of vaccination for yellow fever or with any other live vaccines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Response assessment according to the criteria IMWG | 15-17 month
  compare the Response assessment in both arms: the Very good partial remission rate (according to the criteria IMWG) achieved with four courses of VTD with that achieved with four courses of VCD

SECONDARY OUTCOMES:
Response assessment according to the criteria IMWG | 15 - 17 month
  compare the Response assessment in both arms: the following parameters after induction treatment with four courses of VTD or four courses of VCD the Complete remission rate (according to the criteria IMWG)
Number of Adverse Events | 15-17 month
  To evaluate the Safety of induction therapy
Number of collected stem cell | 17 month
Number of death | 17 month
  To evaluate Overall and Progression-Free Survival
Response assessment according to the criteria IMWG | 15-17 month
  compare the Response assessment in both arms: Compare the following parameters after induction treatment with four courses of VTD or four courses of VCD the Partial remission rate (according to the criteria IMWG)
Number of relapse according to the criteria IMWG | 17 month
  Progression-Free Survival

OTHER OUTCOMES:
Comparison of three techniques for the quantification of urinary monoclonal components in patients with Newly Diagnosed Multiple Myeloma. | 17 month
  The detection and the estimation of the urinary monoclonal components is an inescapable element of the diagnosis and the evaluation of the therapeutic efficacy in the myeloma.
  Urinary protein, electrophoresisin agarose gel is the quantitative method of choice. In these labs, the quantification of the urinary monoclonal peak is not performed. In the absence of quantitative data on urinary monoclonal components, the patient is considered as non-assessable. Recently, the company Sebia has developed the quantification on two other materials used specifically for the characterization of monoclonal component and / or proteinuria (HYDRAGEL BENCE JONES and HYDRAGEL URINE PROFILE).
  The objective of this study is to compare the quantification of monoclonal components between the reference HR electrophoresis technique and the other two above-mentioned techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MOREAU, Principal Investigator — Nantes University Hospital
Locations (63):
- France (63):
  - CHU Angers, Angers, Angers
  - Hôpital Pitié-Salpétrière, Paris, Paris
  - Centre Hospitalier de la région d'Annecy, Annecy, Pringy
  - CHRU Hôpital Sud, Amiens
  - Centre Hospitalier Argenteuil, Argenteuil
  - Centre Hospitalier H.Duffaut, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHRU de Besançon, Besançon
  - Hôpital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre hospitalier Pierre Oudot, Bourgoin
  - Hôpital A.Morvan, Brest
  - CHU Caen Côte de Nacre, Caen
  - CH René Dubos, Cergy-Pontoise
  - Centre Hospitalier William Morey, Chalon/saone
  - Hôpital d'instruction des armées Percy, Clamart
  - CHU d'Estaing, Clermont-Ferrand
  - Hôpitaux civils de Colmar, Colmar
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CHRU Dijon, Dijon
  - Centre Hospitalier Général, Dunkirk
  - CHRU - Hôpital A.Michallon, Grenoble
  - Centre hospitalier départemental Vendée, La Roche-sur-Yon
  - Hôpital Louis Pasteur, Le Coudray
  - Centre Jean Bernard, Le Mans
  - CH Le Mans, Le Mans
  - Hopital Saint Vincent de Paul, Lille
  - CHRU - Hôpital Claude Huriez, Lille
  - CHU de Limoges, Limoges
  - Hôpital Du Scorff, Lorient
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - CHR Metz Thionville, Metz
  - Centre Hospitalier intercommunale Meulan les mureaux, Meulan-en-Yvelines
  - Hopital E Muller, Mulhouse
  - Nantes University Hospital, Nantes
  - Hôpital de l'Archet 1, Nice
  - Groupe Hospitalo-Universitaire Carémeau, Nîmes
  - Institut CURIE, Paris
  - Hôpital Cochin, Paris
  - CHU - Hôpital St-Antoine, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - AP-HP Hôpital Necker, Paris
  - CH Saint Jean, Perpignan
  - CHRU - Hôpital du Haut Lévêque, Pessac
  - Centre Hospitalier de PERIGUEUX, Périgueux
  - Centre Hospitalier Lyon sud, Pierre-Bénite
  - CHRU - Hôpital Jean Bernard, Poitiers
  - Hôpital R.Debré, Reims
  - CHRU - Hôpital de Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Yves le Foll, Saint-Brieuc
  - Centre René Huguenin, Saint-Cloud
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Centre Hospitalier, Saint-Quentin
  - Centre hospitalier, St-Malo
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHRU - Hôpital Purpan, Toulouse
  - CHRU - Hôpital Bretonneau, Tours
  - CHRU - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique Vannes et Auray, Vannes

REFERENCES:
- [Derived] Rosinol L, Hebraud B, Oriol A, Colin AL, Rios Tamayo R, Hulin C, Blanchard MJ, Caillot D, Sureda A, Hernandez MT, Arnulf B, Mateos MV, Macro M, San-Miguel J, Belhadj K, Lahuerta JJ, Garelik MB, Blade J, Moreau P. Integrated analysis of randomized controlled trials evaluating bortezomib + lenalidomide + dexamethasone or bortezomib + thalidomide + dexamethasone induction in transplant-eligible newly diagnosed multiple myeloma. Front Oncol. 2023 Nov 2;13:1197340. doi: 10.3389/fonc.2023.1197340. eCollection 2023. PMID 38023148